CLINICAL TRIAL: NCT02294175
Title: RCT: Larval Debridement Therapy Versus Sharp Debridement to Remove Biofilm From Chronic Lower Extremity or Diabetic Foot Ulcers
Brief Title: Larval Debridement Therapy Versus Sharp Debridement to Remove Biofilm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Florida Foundation for Research and Education (Other)
Collaborators: North Florida/South Georgia Veterans Health System (Other); Biomonde (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201400590
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Lower Extremity or Diabetic Foot Ulcers; Bacterial Infection
Keywords: larva; debridement; lower extremity or diabetic foot ulcer; biofilm; infection; chronic wound
MeSH Terms: conditions — Diabetic Foot; Bacterial Infections; Infections | interventions — Maggot Debridement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Larval Debridement Therapy (Active Comparator): Larval debridement therapy intervention (Biobags) filled with sterile green bottle fly maggots (larvae) placed in open, chronic lower extremity or diabetic foot ulcer once every 4 days for total of 2 applications over the 8 day study period.
  Interventions: Device: Larval Debridement Therapy
- Sharp Debridement Therapy (Active Comparator): Bedside sharp debridement therapy as a comparator performed by wound care clinician once every 7 days in a chronic lower extremity or diabetic foot ulcer for a total of 2 sharp debridements over the 8 day study period.
  Interventions: Procedure: Bedside Sharp Debridement

INTERVENTIONS:
Device: Larval Debridement Therapy — small sterile mesh bags containing live maggots placed into an open chronic wound to remove necrotic tissue and bacterial biofilm
  Other Names: LDT; Maggot Debridement; MDT; Maggots; Medicinal Maggots; Larvae; Biobags
  Arms: Larval Debridement Therapy
Procedure: Bedside Sharp Debridement — The use of a sharp clinical instrument (currette, scalpel, scissors, forceps) by a qualified clinician to remove necrotic tissue and bacterial biofilm from an open chronic wound
  Other Names: Sharp debridement; Sharps
  Arms: Sharp Debridement Therapy

SUMMARY:
This is a prospective study of Veterans with chronic lower extremity or diabetic foot ulcers who will be randomized to either a Larval Debridement Therapy group (Biobags every 4 days x 2 applications) or a Sharp Debridement Therapy group (standard or control weekly x 2) during an 8 day study period.

DETAILED DESCRIPTION:
Drug resistant organisms and bacterial biofilm pose an increasing threat to the health of millions of individuals world-wide. These organisms are being identified with an alarming prevalence among persons with chronic wounds. The presence of necrotic tissue has been associated with the deterioration of open wounds and serves as a breeding ground and nutrient source for bacteria. The removal of necrotic tissue is widely accepted as required for optimal wound healing.

The primary purpose of this study is to assess the efficacy of larval debridement therapy (LDT) with bagged, sterilized, live, medicinal blow fly (Lucilia sericata) larvae (or " BioBags") versus bedside sharp debridement in removing harmful bacteria, biofilm and necrotic tissue from chronic wounds to promote wound healing. Characteristics associated with chronic wound environments will be evaluated through analysis of samples of tissue taken from wound beds before and after both types of debridement. One hundred and forty patients ≥ 21 years of age (and their caregivers and wound providers)with an open, full thickness wound which is healing by secondary intention (of greater than 8 weeks duration and requires debridement) will be invited to participate. This recruitment number accounts for estimated 10% attrition rate, so final sample number is anticipated to be 296 or 128 Veteran subjects (64 in each arm) and 128 caregivers, and 6 providers (and total of 34 subjects which may be lost to follow up). Samples of wound bed tissue and slough tissue (if present) will be collected on Days 0, 4 and 8 or prior to and after each larval debridement intervention or sharp debridement (control). Photos will be taken of the wound bed on Days 0, 4 and 8 or just prior to and after each debridement method. A randomized sampling procedure will place individuals into one of two groups: The intervention group will receive larval debridement therapy once every 4 days for 2 applications (with saline moistened gauze as cover dressing changed daily) and the control group will receive sharp debridement therapy every 7 days for 2 debridements (with wound gel dressing changed daily).

ELIGIBILITY:
Inclusion Criteria:

* Veterans over 21 years of age
* with chronic lower extremity or diabetic foot ulcers (wound duration over 8 weeks)
* who at the clinician's judgment requires wound debridement (25% or more of wound bed covered with non-viable tissue)
* wound size 1.5 cm (roughly the size of a quarter) or larger in diameter

Exclusion Criteria:

* Cognitive impairment that would interfere with patient signing own Informed Consent
* Veterans on active anticoagulant therapy with most recent (within last week) PT/INR (international normalized ratio of prothrombin time) > 3.0, or other significant bleeding risk
* Active immune suppression just prior to or during study (on systemic corticosteroids* within 7 days prior, or chemotherapy for cancer or RA treatment within 4 weeks prior to study, or with diagnosis of HIV/AIDS) - *Nasal steroid sprays will not be excluded
* Active systemic antibiotics is an exclusion
* Absent dorsalis pedis pulses and Ankle Brachial Index (ABI) < 0.5 is an exclusion (indicates critical limb ischemia).
* Other possible reasons participants could be removed from this study include: transfers to other non-VA facilities, participant is unable to tolerate tissue sampling even with local anesthesia, and/or inability to comply with scheduled research visits. Furthermore, if the participant has significant wound healing so that sampling is not possible after the initial sampling, they will be removed from the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2018-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Cowan, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (2):
- United States (2):
  - North Florida Regional Medical Center, Gainesville, Florida
  - North Florida / South Georgia Veterans Health System, Gainesville, Florida

REFERENCES:
- [Derived] Sen CK, Roy S, Mathew-Steiner SS, Gordillo GM. Biofilm Management in Wound Care. Plast Reconstr Surg. 2021 Aug 1;148(2):275e-288e. doi: 10.1097/PRS.0000000000008142. PMID 34398099

RESULTS

PARTICIPANT FLOW:
Groups:
- Larval Debridement Therapy (LDT) - Patients: Larval debridement therapy intervention (Biobags) filled with sterile green bottle fly maggots (larvae) placed in open, chronic lower extremity or diabetic foot ulcer once every 4 days for total of 2 applications over the 8 day study period.
  Larval Debridement Therapy: small sterile mesh bags containing live maggots placed into an open chronic wound to remove necrotic tissue and bacterial biofilm
- Sharp Debridement Therapy (SDT) - Patients: Bedside sharp debridement therapy as a comparator performed by wound care clinician once every 7 days in a chronic lower extremity or diabetic foot ulcer for a total of 2 sharp debridements over the 8 day study period.
  Bedside Sharp Debridement: The use of a sharp clinical instrument (currette, scalpel, scissors, forceps) by a qualified clinician to remove necrotic tissue and bacterial biofilm from an open chronic wound
Period: Overall Study
Arm/Group | Larval Debridement Therapy (LDT) - Patients | Sharp Debridement Therapy (SDT) - Patients
Started | 23 | 22
Completed | 18 | 16
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 1 | 2
Not completed — pt taking excluded medication | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — wound healed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (8.5) | 64.9 (6.6) | 65.4 (7.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 16 | 13 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 3 | 4 | 7
  Hispanic/Latino | 0 | 1 | 1
  White/Caucasian | 11 | 11 | 22
  Other | 1 | 0 | 1
  Not documented | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 16 | 34
Current Smokers [Count of Participants; unit: Participants] | 3 | 5 | 8
History of wounds [Count of Participants; unit: Participants]
  History of diabetic lower extremity wounds | 10 | 11 | 21
  Venous leg ulcers | 4 | 3 | 7
  Other lower extremity wounds | 2 | 2 | 4
  None documented | 2 | 0 | 2
Marital/partner status [Count of Participants; unit: Participants]
  Married/partner | 7 | 7 | 14
  Single | 8 | 9 | 17
  Widow/Widower | 1 | 0 | 1
  Declined to answer | 2 | 0 | 2
Suspected duration of wound at enrollment [Count of Participants; unit: Participants]
  Over 8 weeks unknown total duration | 2 | 1 | 3
  Over 8 weeks but under 6 months duration | 2 | 5 | 7
  Over 6 months but under 1 year duration | 7 | 2 | 9
  One year or longer duration | 5 | 8 | 13
  Not documented | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Total Bacteria Colony Forming Units (CFUs; Natural-log Transformed), With Tryptic Soy Agar (TSA) Plating
Description: Differences in total bacterial colony forming units (CFUs) between LDT and SDT arms at Day 0, with Tryptic Soy Agar (TSA) plating. Raw outcomes were natural-log transformed due to skewed distribution. Higher scores correspond to a greater number of bacterial CFUs (i.e., worse outcome).
Time Frame: Day 0 (Baseline), Day 4, Day 8
Population: Statistical analysis was performed on a subset of participants (n=32) due to missing data on one or more days of measurement.
Measure: Mean (Standard Deviation); unit: Natural Log Transformed Bacterial CFU
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy
Number analyzed (Participants) | 17 | 15
Natural Log Transformed Bacterial CFU
  Day 0 | 9.6561 (3.10402) | 9.6880 (1.75013)
  Day 4 | 11.9611 (1.68800) | 9.1547 (2.57417)
  Day 8 | 11.4864 (2.05378) | 10.4479 (2.25869)
Statistical Analysis 1: Comparison: Larval Debridement Therapy vs Sharp Debridement Therapy; Repeated Measures Analysis of Variance (RMANOVA) to test for effects of treatment arm, time, and treatment-by-time interaction. The effect of interest is the treatment-by-time interaction, i.e, whether the reduction of bacterial CFUs over time varies according to treatment arm; Test type: Superiority; p = .029, Repeated Measures ANOVA — Repeated Measures ANOVA. The interaction effect is controlling for any potential main effects of treatment arm (SDT vs LDT) and time (days 0, 4, 8); Greenhouse-Geisser corrections were applied to the F test degrees of freedom due to violation of the sphericity assumption (p<.05 for Mauchly's W)

2. Primary Outcome: Total Bacteria Colony Forming Units (CFUs; Natural-log Transformed), With MacConkey Agar Plating
Description: Differences in total bacterial colony forming units (CFUs) between LDT and SDT arms at Day 0, with MacConkey Agar plating. Raw outcomes were natural-log transformed due to skewed distribution. Higher scores correspond to a greater number of bacterial CFUs (i.e., worse outcome).
Time Frame: Day 0 (Baseline), Day 4, Day 8
Population: Statistical analysis was performed on a subset of participants (n=33) due to missing data on one or more days of measurement.
Measure: Mean (Standard Deviation); unit: Natural Log Transformed Bacterial CFU
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy
Number analyzed (Participants) | 18 | 15
Natural Log Transformed Bacterial CFU
  Day 0 | 4.5512 (4.32429) | 5.4009 (4.76243)
  Day 4 | 8.9408 (3.64582) | 6.2482 (4.32648)
  Day 8 | 8.9198 (4.33985) | 6.8660 (4.80509)
Statistical Analysis 1: Comparison: Larval Debridement Therapy vs Sharp Debridement Therapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .037, Repeated Measures ANOVA — Repeated Measures ANOVA. This interaction effect is controlling for any potential main effects of treatment arm (SDT vs LDT) and time (days 0, 4, 8); [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Total Bacteria Colony Forming Units (CFUs; Natural-log Transformed),With Phenylethyl Alcohol (PEA) Plating
Description: Differences in total bacterial colony forming units (CFUs) between LDT and SDT arms at Day 0, with Phenylethyl Alcohol (PEA) plating. Raw outcomes were natural-log transformed due to skewed distribution. Higher scores correspond to a greater number of bacterial CFUs (i.e., worse outcome).
Time Frame: Day 0 (Baseline), Day 4, Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Natural Log Transformed Bacterial CFU
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy
Number analyzed (Participants) | 18 | 15
Natural Log Transformed Bacterial CFU
  Day 0 | 7.0633 (4.45210) | 8.7514 (1.56580)
  Day 4 | 9.8704 (2.69279) | 8.5673 (2.64319)
  Day 8 | 9.2877 (2.71007) | 9.7341 (2.52994)
Statistical Analysis 1: Comparison: Larval Debridement Therapy vs Sharp Debridement Therapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .012, Repeated Measures ANOVA — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Reviewer Assessment of Visible Wound Improvement
Description: For each patient, wound photos were taken at days 0, 4, and 8 and given to wound specialists. Wound specialists reviewed photos to assess whether there was visible reduction in amount of necrotic or non-viable tissue remaining in the wound bed at day 8--i.e., whether the wound appeared to be improved (yes vs. no). The percentage of reviewers (out of 4) who responded "yes" that the wound appeared improved was calculated for each patient. Thus, each patient received a score for percentage of reviewers who saw visual improvement; the means and standard deviations for these percentages were compared between LDT and SDT groups. Higher scores correspond to better outcomes (higher proportion of reviewers who responded that wounds appeared visibly improved).
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: percentage of reviewers
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy
Number analyzed (Participants) | 18 | 16
percentage of reviewers | 61.11 (39.503) | 71.88 (32.755)
Statistical Analysis 1: Comparison: Larval Debridement Therapy vs Sharp Debridement Therapy; Test type: Superiority; p = .397, t-test, 2 sided

5. Secondary Outcome: Inflammatory Biomarker MMP-9
Description: Using Enzyme Linked Immunosprbent Assay (ELISA), the levels of active Matrix Metalloproteinase type 9 (MMP-9) was calculated and expressed as pg/ml of wound fluid and pg/mg protein. Raw outcomes were natural-log transformed due to skewed distribution. Higher scores indicate worse outcomes.
Time Frame: Day 0 (Baseline), Day 4, Day 8
Population: Statistical analysis was performed on a subset of participants (n=20) due to missing data on one or more days of measurement.
Measure: Mean (Standard Deviation); unit: Natural Log Transformed MMP-9 in pg/ml
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy
Number analyzed (Participants) | 11 | 9
Natural Log Transformed MMP-9 in pg/ml
  Day 0 | 2.8538 (0.83493) | 2.8965 (0.87010)
  Day 4 | 2.7847 (0.76985) | 2.7260 (0.71122)
  Day 8 | 2.9985 (0.63257) | 2.6861 (0.84722)
Statistical Analysis 1: Comparison: Larval Debridement Therapy vs Sharp Debridement Therapy; Repeated Measures Analysis of Variance (RMANOVA) to test for effects of treatment arm, time, and treatment-by-time interaction. The effect of interest is the treatment-by-time interaction, i.e, whether change in MMP-9 over time varies according to treatment arm; Test type: Superiority; p = .661, Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Inflammatory Biomarker IL6
Description: The levels of active IL6 was calculated using Enzyme Linked Immunosprbent Assay (ELISA) and reported in ng/ml. Raw outcomes were natural-log transformed due to skewed distribution. Higher scores indicate worse outcomes.
Time Frame: Day 0 (Baseline), Day 4, Day 8
Population: Statistical analysis was performed on a subset of participants (n=27) due to missing data on one or more days of measurement.
Measure: Mean (Standard Deviation); unit: Natural Log Transformed IL6 in ng/ml
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy
Number analyzed (Participants) | 15 | 12
Natural Log Transformed IL6 in ng/ml
  Day 0 | 3.4889 (1.29396) | 3.5748 (1.94347)
  Day 4 | 4.2287 (1.65271) | 4.2233 (1.18058)
  Day 8 | 4.0069 (1.37460) | 4.0096 (1.68661)
Statistical Analysis 1: Comparison: Larval Debridement Therapy vs Sharp Debridement Therapy; Repeated Measures Analysis of Variance (RMANOVA) to test for effects of treatment arm, time, and treatment-by-time interaction. The effect of interest is the treatment-by-time interaction, i.e, whether change in IL6 over time varies according to treatment arm; Test type: Superiority; p = .979, Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Satisfaction With Debridement: Overall Satisfaction With Method, Day 8
Description: Satisfaction (Overall) item score. This item is from a Satisfaction with Debridement survey, designed to measure satisfaction with debridement method, aesthetic questions regarding debridement, ease of use/care, and wound pain. Individual item scores range from 0 to 10, with higher scores indicating better outcomes (higher overall satisfaction).
Time Frame: Day 8
Population: Statistical analysis was performed on a subset of participants (n=30) due to missing data on one or more measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy
Number analyzed (Participants) | 15 | 15
score on a scale | 7.27 (3.642) | 7.13 (3.642)
Statistical Analysis 1: Comparison: Larval Debridement Therapy vs Sharp Debridement Therapy; Kolmogorov-Smirnov Z test was used as a non-parametric test to compare rank scores between treatment arms (similar to Mann-Whitney, but potentially more powerful); Test type: Superiority; p = .999, Kolmogorov-Smirnov Z

8. Secondary Outcome: Satisfaction: Aesthetic Unpleasantness of Debridement, Day 8
Description: Survey item score for Aesthetic Unpleasantness of debridement. This item is from a Satisfaction with Debridement survey. Individual item scores range from 0 to 10, with higher scores on the aesthetic unpleasantness item indicating worse outcomes
Time Frame: Day 8
Population: Statistical analysis was performed on a subset of participants (n=32) due to missing data on one or more measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy
Number analyzed (Participants) | 16 | 16
score on a scale | 2.63 (2.872) | 3.75 (4.266)
Statistical Analysis 1: Comparison: Larval Debridement Therapy vs Sharp Debridement Therapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .415, Kolmogorov-Smirnov Z

9. Secondary Outcome: Satisfaction: Difficulty of Use/Care, Day 8
Description: Survey item score for Difficulty of Use/Care of debridement. This item is from a Satisfaction with Debridement survey. Individual item scores range from 0 to 10, with higher scores on the difficulty item indicating worse outcome (higher difficulty of use/care for debridement method).
Time Frame: Day 8
Population: Statistical analysis was performed on a subset of participants (n=31) due to missing data on one or more measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy
Number analyzed (Participants) | 15 | 16
score on a scale | 1.60 (2.530) | 1.88 (3.243)
Statistical Analysis 1: Comparison: Larval Debridement Therapy vs Sharp Debridement Therapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .993, Kolmogorov-Smirnov Z

10. Secondary Outcome: Satisfaction: Wound Pain, Day 8
Description: Satisfaction survey to measure satisfaction with debridement method, aesthetic questions regarding debridement, ease of use/care, and wound pain. Pain was measured using the Defense and Veterans Pain Rating Scale (DVPRS). Individual item scores range from 0 to 10, with higher scores on the DVPRS indicating higher pain and worse outcomes.
Time Frame: Day 8
Population: Statistical analysis was performed on a subset of participants (n=30) due to missing data on one or more measures.
Measure: Mean (Standard Deviation); unit: DVPRS (Pain) Score
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy
Number analyzed (Participants) | 14 | 16
DVPRS (Pain) Score | 4.14 (3.110) | 3.63 (3.284)
Statistical Analysis 1: Comparison: Larval Debridement Therapy vs Sharp Debridement Therapy; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = .990, Kolmogorov-Smirnov Z

ADVERSE EVENTS:
Time Frame: period of time over which adverse event data were collected was 3 years (11/25/2014 to 11/25/2017).
Description: definitions were not different, any adverse event reported by participant, clinician, or study team were recorded and reported to IRB as per regulatory protocol
Arm/Group | Larval Debridement Therapy | Sharp Debridement Therapy
All-Cause Mortality (participants affected / at risk) | 1/18 | 1/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

LIMITATIONS AND CAVEATS:
This study was underpowered to observe significant difference between SDT and LDT groups. Aversion to LDT we anticipated in subjects, caregivers, and clinicians were not encountered. Almost all subjects in SDT group elected to try LDT after study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT02294175/Prot_SAP_000.pdf